CLINICAL TRIAL: NCT02490150
Title: Administration of Corifollitropin Alfa on Day 5 Versus Day 7 After Last Oral Contraceptive Pill in a GnRH (Gonadotropin-releasing Hormone ) Antagonist Protocol in Donors
Brief Title: Corifollitropin Alfa on D5 Versus D7 After Contraceptive Pill
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Collaborators: Francisca Martínez (Unknown); Buenaventura Coroleu (Unknown); Elisabet Clua (Unknown); Ignacio Rodríguez (Unknown)
Responsible Party: Principal Investigator, Ignacio Rodriguez, MD., Fundacion Dexeus
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDQ-COR-2014-01
Record Dates: First submitted 2015-06-22; First posted 2015-07-03 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Oocyte Donation
Keywords: Corifollitropin alfa; Stimulation protocol
MeSH Terms: interventions — follicle stimulating hormone, human, with HCG C-terminal peptide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day 5 (Experimental): Administration of corifollitropin alfa on Day 5 after last oral contraceptive pill in a GnRH antagonist protocol in donors.
  Interventions: Drug: Corifollitropin alfa
- Day 7 (Active Comparator): Administration of corifollitropin alfa on Day 7 after last oral contraceptive pill in a GnRH antagonist protocol in donors.
  Interventions: Drug: Corifollitropin alfa

INTERVENTIONS:
Drug: Corifollitropin alfa

SUMMARY:
To evaluate if the administration of corifollitropin alfa on day 7 instead of on day 5 after pre-treatment with oral contraceptive pill results in a reduced total rFSH (recombinant follicle stimulating hormone ) consumption in a GnRH antagonist protocol in donors.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-35 y old ,with regular spontaneous menstrual cycles of 25-30 days length
* Who had vaginal sexual intercourse or have no inconvenient for vaginal explorations
* Donors can´t have more than 6 children (neither own or after donations)
* Not be adopted or being born after a gamete donation pregnancy
* BMI between 18-28 kg/m2
* Height > 1.55cm
* Gynecological and general examination with Pap smear, HIV, HCV (hepatitis C virus ), HBV (hepatitis B virus ) and RPR(rapid plasma reagin test ) negative serology, and with normal karyotype
* No abnormal Psychological profile
* Discard any disease: blood disorders, neurodegenerative/psychiatric diseases, Fragile X Syndrome, cystic fibrosis carrier, oncology diseases.
* Without psychological/psychiatric family history
* Will conform to the protocol for the duration of the study
* Willingness of adhesion to protocol during the whole study period
* Signed informed consent

Exclusion Criteria:

* Polycystic ovarian syndrome
* Antral follicle count > 20
* Hypersensitivity to the active substance or any of the excipients
* Abnormal vaginal bleeding of unknown ethiology
* Presence of ovarian cysts or increased size ovaries
* History of ovarian hyperstimulation syndrome
* Previous controlled ovarian stimulation cycle with more than 30 follicles ≥ 11mm
* Previous abdominal surgery that contraindicated the practice of follicular puncture
* HIV, HCV, HBV positive serology in women or partner
* Important systemic diseases that could interfere with gonadotrophin treatment (ovarian and hypothalamic tumors…)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
total dosis of rFSH (IU) | donors will be followed until the end of stimulation period, an expected average of 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Quiron Dexeus, Barcelona, Spain

REFERENCES:
- [Background] Blockeel C, Polyzos NP, Derksen L, De Brucker M, Vloeberghs V, van de Vijver A, De Vos M, Tournaye H. Administration of corifollitropin alfa on Day 2 versus Day 4 of the cycle in a GnRH antagonist protocol: a randomized controlled pilot study. Hum Reprod. 2014 Jul;29(7):1500-7. doi: 10.1093/humrep/deu105. Epub 2014 May 9. PMID 24813196